CLINICAL TRIAL: NCT06784037
Title: Optimal Positive End-Expiratory Pressure in Robotic-Assisted Thoracic Surgery Without Capnothorax
Status: Enrolling by invitation | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Other Study IDs: HCB/2024/0103
Record Dates: First submitted 2024-12-16; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-12

CONDITIONS: Robotic Thoracic Surgery; Mechanical Ventilation; Positive End Expiratory Pressure (PEEP)
Keywords: robotic lung surgery; PEEP; capnothorax

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- URATS: Robotic lung surgery with no capnothorax: Uniportal robotic lung resection under no capnothorax

SUMMARY:
The aim of this study is to assess the impact on lung mechanics during robotic lung resection when no capnothorax is used.

DETAILED DESCRIPTION:
Assess the improvement of oxygenation, ventilation and lung mechanics in patients ventilated with individualized PEEP without capnothorax. PEEP requirement and lung mechanics without capnothorax will be compared with a historical cohort population of robotic surgery with capnothorax.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing uniportal robotic lung resection under no capnothorax

Exclusion Criteria:

* Refusal to participate
* Contraindications to recruitment maneuvers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving uniportal robotic assisted lung resection with no capnothorax
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Respiratory airway pressures | During intra-operative mechanical ventilation (4 hours)
  Respiratory airway pressures (peak pressure, plateau pressure and PEEP in cmH2O)
Respiratory rate | During intra-operative mechanical ventilation (4 hours)
  Respiratory rate (in cycles per minute)
Respiratory system compliance | During intra-operative mechanical ventilation (4 hours)
  Respiratory pressures measurement will be combined to obtain respiratory system compliance.
  Respiratory system compliance = (plateau pressure-PEEP) / respiratory tidal volume (expressed in cmH2O/mL)

SECONDARY OUTCOMES:
Arterial blood gas parameters: pO2 | During intra-operative mechanical ventilation (4 hours)
  pO2 in mmHg in arterial blood gas sample
Arterial blood gas parameters: pCO2 | During intra-operative mechanical ventilation (4 hours)
  pCO2 in mmHg in arterial blood gas sample
Arterial blood gas parameters: pH | During intra-operative mechanical ventilation (4 hours)
  pH of arterial blood gas samples (no unit can be applied)
Arterial blood gas parameters: sodium bicarbonate | During intra-operative mechanical ventilation (4 hours)
  Arterial blood sample sodium bicarbonate concentration (in mmol/L)
Arterial blood gas parameters: base excess | During intra-operative mechanical ventilation (4 hours)
  Base excess in arterial blood gas samples in mEq/L

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic Barcelona, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided